CLINICAL TRIAL: NCT01453023
Title: A Randomized, Double-blind, Repeat Dose, Two Period Crossover Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Inhaled Fluticasone Furoate/Vilanterol 100/25 Micrograms in Children Aged 5 to 11 Years With Persistent Asthma
Brief Title: Inhaled Fluticasone Furoate/Vilanterol Safety and Tolerability, PK and PD Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 112777
Record Dates: First submitted 2011-10-06; First posted 2011-10-17 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: pediatric ages 5 to 11 years
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate (Active Comparator): One of two study treatments subjects will receive. Given to allow comparison of FF exposure in combination versus as mono therapy.
  Interventions: Drug: Fluticasone Furoate
- Fluticasone Furoate/Vilanterol (Experimental): One of two study treatments subjects will receive. FF/VI combined is being tested and compared to fluticasone furoate.
  Interventions: Drug: Fluticasone Furoate/Vilanterol

INTERVENTIONS:
Drug: Fluticasone Furoate — 100mcg delivered via a novel dry powder inhaler on days 1-14 of one study treatment period.
  Other Names: FF
  Arms: Fluticasone Furoate
Drug: Fluticasone Furoate/Vilanterol — 100/25 mcg delivered via a novel dry powder inhaler on days 1-14 of one study treatment period.
  Other Names: FF/VI
  Arms: Fluticasone Furoate/Vilanterol

SUMMARY:
This study will investigate the safety and tolerability, pharmacokinetics, and pharmacodynamics of fluticasone furoate/vilanterol (FF/VI) 100/25mcg administered using the novel dry powder inhaler in children aged 5 to 11 years with persistent asthma.

DETAILED DESCRIPTION:
This study will investigate the safety and tolerability, pharmacokinetics, and pharmacodynamics of fluticasone furoate/vilanterol (FF/VI) 100/25mcg administered using the novel dry powder inhaler in children aged 5 to 11 years with persistent asthma. Fluticasone furoate (FF, GW685698) is a novel once daily inhaled corticosteroid (ICS) and vilanterol (VI, GW642444) is an inhaled once daily long-acting beta2 agonist (LABA). FF/VI is a novel ICS/LABA combination with once-daily dosing being developed for the treatment of asthma in adults, adolescents, and children of 5 years and above.

This study will be a randomized, double-blind, repeat dose, two period crossover study, with FF as the control. During each of two treatment periods subjects will receive either FF/VI 100/25 micrograms (mcg) or FF 100 mcg daily on 14 consecutive mornings via the novel dry powder inhaler. Approximately 26 subjects will be recruited into this study, with a target of 20 completed subjects. Safety, tolerability, pharmacokinetics and glucose , potassium and cortisol levels will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a study physician, based medical history, physical examination, laboratory testing, and electrocardiogram (ECG); with no significant medical condition apart from asthma, eczema, or rhinitis. A subject with a clinical abnormality or laboratory parameters outside the reference range for this study may be included if the Investigator and GSK Medical Monitor agree the finding is unlikely to introduce additional risk factors or interfere with the study procedures.
* Male and pre-menarchial female subjects aged 5 to less than 12 years on the last planned treatment day are eligible for this study. Pre-menarchial females are defined as any female who has not begun menses and is considered Tanner Stage 2 or less.
* Diagnosis of asthma at least 6 months prior to screening.
* Stable asthma therapy (fluticasone propionate, total daily dose less than or equal to 400 microgram or equivalent) and short acting beta-agonist (SABA) inhaler for at least 4 weeks prior to screening.
* Subjects must be controlled on their existing asthma treatment at screening, which will be continued during the run-in, washout and run-out periods (but not during active treatment periods). Control is defined as a Childhood Asthma Control Test score of >19 and (Peak Expiratory Flow) PEF more than 75 percent predicted.
* Subjects must demonstrate an ability to accept and effectively use a demonstration inhaler from the demonstration kits provided.
* Subjects must weigh at least 20 kilograms.
* The subject and parent/guardian are able to understand and comply with protocol requirements, instructions, and protocol stated restrictions. The parent or guardian must have the ability to read, write, and record diary information collected throughout the study. The parent or guardian must have the ability to manage study drug administration and PEF assessments.
* At least one parent/guardian has signed and dated the written informed consent prior to admission to the study. This will be accompanied by informed assent from the subject for children aged 7 to 11 years.

Exclusion Criteria:

* Subjects with a history of life-threatening asthma, an asthma exacerbation requiring systemic corticosteroids or Emergency Room attendance (within 3 months) or requiring hospitalization (within 6 months) prior to screening.
* Subjects with any medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear, not resolved within 4 weeks of screening leading to a change in asthma management; or, in the opinion of the investigator, is likely to affect the subject's asthma status or ability to participate in the study.
* Clinical visual evidence of oral candidiasis at screening.
* Subjects currently receiving (or have received within 4 weeks of screening) asthma therapies including theophyllines, long-acting inhaled beta-agonists, oral beta-agonists, or who have changed their asthma medication within 4 weeks of screening.
* Significant abnormality of rate, interval, conduction or rhythm in the 12-lead ECG (electrocardiogram), determined by the investigator in conjunction with the age and gender of the child and the assessment provided by the remote analysis service.
* QTcF (QT interval corrected for heart rate using Fridericia's formula) more than 450 milliseconds or an ECG not suitable for QT measurement (e.g. poorly defined termination of the T wave).
* Aspartarte aminotransferase, Alanine aminotransferase, alkaline phosphatase and bilirubin more than 1.5 times Upper Limit of Normal (ULN) (isolated bilirubin more than 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percent).
* A known or suspected sensitivity to any constituents of the novel dry powder inhaler (i.e. lactose or magnesium stearate) (e.g. history of severe milk protein allergy)
* Any adverse reaction including immediate or delayed hypersensitivity to any beta-2-agonist, sympathomimetic drug, or any intranasal, inhaled or systemic corticosteroid therapy.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of the lesser of 50 millilitres (mL) or 3mL per kilogram within a 56 day period.
* Parent/guardian has a history of psychiatric disease, intellectual deficiency, substance abuse, or other condition (e.g. inability to read, comprehend and write) which will limit the validity of consent to participate in this study.
* Unwillingness or inability of the subject or parent/guardian to follow the procedures outlined in the protocol.
* Subject who is mentally or legally incapacitated.
* Children who are wards of the state or government.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Huntington Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112777 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into one of two cohorts based upon age; the younger cohort was enrolled after a review of the safety/pharmacokinetic data of at least six participants from the older cohort. Each participant was assigned to treatment randomly; assignment was not to be influenced by whether participants were in Cohort 1 or Cohort 2.
Pre-assignment Details: A Baseline assessment was carried out on Day 1 of the first treatment period. Participants were then randomized to one of the two possible treatments fluticasone furoate [FF] 100 µg/Vilanterol [VI] 25 µg.or FF 100 µg, followed by a cross over after a washout period of at least 7 days.
Groups:
- FF 100 µg/VI 25 µg in TP 1 and FF 100 µg in TP 2: Participants received fluticasone furoate (FF) 100 micrograms (µg)/Vilanterol (VI) 25 µg in Treatment Period 1 and FF 100 µg in Treatment Period 2. The first 14-day treatment period was followed by a washout period of at least 7 days. Inhaled FF 100 µg/VI 25 µg and FF 100 µg were administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler.
- FF 100 µg in TP 1 and FF 100 µg/VI 25 µg in TP 2: Participants received FF 100 µg in Treatment Period 1 and FF 100 µg/VI 25 µg in Treatment Period 2. The first 14-day treatment period was followed by a washout period of at least 7 days. Inhaled FF 100 µg/VI 25 µg and FF 100 µg were administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler.
Period: Treatment Period (TP) 1
Arm/Group | FF 100 µg/VI 25 µg in TP 1 and FF 100 µg in TP 2 | FF 100 µg in TP 1 and FF 100 µg/VI 25 µg in TP 2
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Met Protocol-defined Stopping Criteria | 0 | 1
Period: Washout Period
Arm/Group | FF 100 µg/VI 25 µg in TP 1 and FF 100 µg in TP 2 | FF 100 µg in TP 1 and FF 100 µg/VI 25 µg in TP 2
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | FF 100 µg/VI 25 µg in TP 1 and FF 100 µg in TP 2 | FF 100 µg in TP 1 and FF 100 µg/VI 25 µg in TP 2
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FF 100 µg/VI 25 µg and FF 100 µg in TPs 1 and 2: All participants who received FF 100 µg/VI 25 µg in Treatment Period 1 and FF 100 µg in Treatment Period 2 or FF 100 µg in Treatment Period 1 and FF 100 µg/VI 25 µg in Treatment Period 2. The first 14-day treatment period was followed by a washout period of at least 7 days. Inhaled FF 100 µg/VI 25 µg and FF 100 µg were administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler.
Arm/Group | FF 100 µg/VI 25 µg and FF 100 µg in TPs 1 and 2
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.1 (1.97)
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3
  White - Arabic/North African Heritage | 1
  White - White/Caucasian/European Heritage | 21
  African American/African Heritage & White | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of study medication until Week 11 (Visit 9)/Early Withdrawal
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: Participants
Groups:
- FF 100 µg/VI 25 µg: Participants received FF 100 µg/VI 25 µg in one of the two 14-day treatment periods. FF 100 µg/VI 25 µg was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
- FF 100 µg: Participants received FF 100 µg in one of the two 14-day treatment periods. FF 100 µg was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Participants
  Any AE | 4 | 1
  Any SAE | 0 | 0

2. Primary Outcome: Basophil, Eosinophil, Lymphocyte, Monocyte, Total Neutrophil, Platelet, and White Blood Cell Count Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelets, and white blood cell (WBC) count at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
10^9 cells per liter (GI/L)
  Basophils, n=21, 23 | 0.025 (0.0175) | 0.025 (0.0153)
  Eosinophils, n=21, 23 | 0.296 (0.3395) | 0.293 (0.3957)
  Lymphocytes, n=21, 23 | 2.062 (0.8462) | 2.339 (0.7391)
  Monocytes, n=21, 23 | 0.244 (0.1188) | 0.222 (0.1375)
  Total neutrophils, n=21, 23 | 3.805 (2.4090) | 3.106 (1.3526)
  Platelets, n=21, 23 | 270.5 (92.27) | 299.0 (73.66)
  WBC count, n=21, 23 | 6.43 (2.889) | 5.98 (1.897)

3. Primary Outcome: Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of hemoglobin and MCHC at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Grams per liter (g/L)
  Hemoglobin, n=21, 23 | 125.9 (13.49) | 128.0 (6.52)
  MCHC, n=21, 23 | 330.3 (5.83) | 330.8 (7.88)

4. Primary Outcome: Reticulocyte and Red Blood Cell (RBC) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of reticulocytes and RBCs at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
10^12 cells per liter (TI/L)
  Reticulocytes, n=21, 23 | 0.07220 (0.037473) | 0.07323 (0.032203)
  RBCs, n=21, 23 | 4.33 (0.467) | 4.38 (0.199)

5. Primary Outcome: Hematocrit Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of hematocrit at Day 14 of the respective treatment period. Hematocrit is a measure of the percentage of the volume of the whole blood that is composed of red blood cells, as determined by separation of red blood cells from the plasma (usually by centrifugation).
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: proportion of 1
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 21 | 23
proportion of 1 | 0.3816 (0.04199) | 0.3866 (0.02160)

6. Primary Outcome: Mean Corpuscle Volume (MCV) Value at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of MCV at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^15 femtoliters (fL) per cell
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 21 | 23
10^15 femtoliters (fL) per cell | 87.9 (2.61) | 88.6 (3.37)

7. Primary Outcome: Mean Corpuscle Hemoglobin (MCH) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of MCH at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 picograms (pg) per cell
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 21 | 23
10^12 picograms (pg) per cell | 29.03 (0.941) | 29.25 (1.116)

8. Primary Outcome: Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), and Gamma Glutamyl Transferase (GGT) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of ALT, ALP, AST, and GGT at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
International units per liter (IU/L)
  ALT, n=22, 24 | 16.9 (14.63) | 17.7 (14.88)
  ALP, n=22, 24 | 278.4 (110.01) | 272.6 (119.48)
  AST, n=22, 24 | 28.2 (8.38) | 29.0 (7.51)
  GGT, n=22, 24 | 14.6 (7.74) | 16.1 (10.36)

9. Primary Outcome: Albumin and Total Protein Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of albumin and total protein at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population, Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Grams per liter
  Albumin, n=22, 24 | 45.5 (1.97) | 45.6 (2.20)
  Total protein, n=22, 24 | 70.4 (2.99) | 70.4 (3.12)

10. Primary Outcome: Calcium, Chloride, Carbon Dioxide (CO2) Content/Bicarbonate, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of calcium, chloride, carbon dioxide content/bicarbonate (CO2/BI), glucose, potassium, sodium, and urea/BUN at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Millimoles per liter (mmol/L)
  Calcium, n=22, 24 | 2.416 (0.0591) | 2.415 (0.0749)
  Chloride, n=22, 24 | 103.3 (1.75) | 103.8 (1.79)
  CO2 content/bicarbonate, n=22, 24 | 19.0 (1.85) | 19.1 (2.05)
  Glucose, n=22, 24 | 4.50 (0.689) | 4.53 (0.523)
  Potassium, n=22, 24 | 4.24 (0.184) | 4.27 (0.265)
  Sodium, n=22, 24 | 138.6 (1.84) | 139.0 (1.85)
  Urea/BUN, n=22, 24 | 4.52 (1.006) | 4.52 (1.108)

11. Primary Outcome: Total Bilirubin, Direct Bilirubin, Creatinine, and Uric Acid Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of total bilirubin, direct bilirubin, creatinine, and uric acid at Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Micromoles per liter (µmol/L)
  Total bilirubin, n=22, 24 | 6.1 (1.44) | 5.9 (1.72)
  Direct bilirubin, n=22, 24 | 1.7 (0.70) | 1.9 (0.41)
  Creatinine, n=22, 24 | 36.00 (7.617) | 37.09 (6.225)
  Uric acid, n=22, 24 | 231.8 (64.85) | 233.8 (54.04)

12. Primary Outcome: Peak Expiratory Flow on Day 1 and Day 14 of the Respective Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF is calculated as the maximum of three readings taken at each timepoint for each participant. Baseline is defined as the maximum pre-dose measurement at Day 1 for each period.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
liters/minute
  Day 1, Baseline, n=25, 25 | 219.0 (53.27) | 223.6 (56.91)
  Day 1, 10 minutes post-dose, n=25, 25 | 218.8 (53.02) | 223.0 (55.15)
  Day 1, 20 minutes post-dose, n=25, 25 | 222.4 (53.50) | 228.2 (56.73)
  Day 1, 1 hour post-dose, n=25, 25 | 223.2 (54.23) | 227.2 (54.07)
  Day 1, 2 hours post-dose, n=25, 25 | 227.0 (55.94) | 228.6 (54.17)
  Day 14, Pre-dose, n=23, 24 | 224.8 (52.86) | 215.0 (50.71)
  Day 14, 20 minutes post-dose, n=23, 24 | 227.2 (52.18) | 218.1 (52.12)
  Day 14, 2 hours post-dose, n=23, 24 | 235.7 (53.16) | 225.8 (48.78)
  Day 14, 12 hours post-dose, n=23, 24 | 238.9 (55.84) | 230.4 (52.54)

13. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Day 1 and Day 14 of the Respective Treatment Period
Description: SBP and DBP were measured at Day 1 and Day 14 of the respective treatment period. Baseline is defined as the pre-dose measurement at Day 1. Change from Baseline was calculated as the Day 14 value minus the Baseline value.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Millimeters of mercury (mmHg)
  Day 1 SBP, Baseline, n=25, 25 | 97.2 (5.41) | 99.9 (6.71)
  Day 1 SBP, 20 minutes, n=25, 25 | -0.1 (2.98) | -0.1 (4.66)
  Day 1 SBP, 1 hour, n=25, 25 | 0.5 (2.87) | 0.4 (3.70)
  Day 1 SBP, 2 hours, n=25, 25 | 0.9 (3.05) | 1.3 (2.95)
  Day 14 SBP, Pre-dose, n=23, 24 | 1.3 (4.32) | -1.2 (6.92)
  Day 14 SBP, 20 minutes, n=23, 24 | 1.3 (4.61) | -1.2 (6.03)
  Day 14 SBP, 1 hour, n=23, 24 | 1.0 (4.42) | -0.8 (6.36)
  Day 14 SBP, 2 hours, n=23, 24 | 1.7 (4.17) | -0.8 (6.34)
  Day 14 SBP, 4 hours, n=23, 24 | 2.1 (4.22) | 0.1 (6.47)
  Day 14 SBP, 8 hours, n=23, 24 | 2.0 (4.33) | -0.4 (7.17)
  Day 1 DBP, Baseline, n=25, 25 | 62.3 (3.54) | 63.6 (3.86)
  Day 1 DBP, 20 minutes, n=25, 25 | 0.3 (2.81) | -0.3 (3.76)
  Day 1 DBP, 1 hour, n=25, 25 | 1.0 (3.17) | 0.8 (3.11)
  Day 1 DBP, 2 hours, n=25, 25 | 0.9 (3.42) | 1.0 (3.38)
  Day 14 DBP, Pre-dose, n=23, 24 | 0.6 (3.54) | 0.2 (3.29)
  Day 14 DBP, 20 minutes, n=23, 24 | 0.1 (3.69) | 0.1 (2.62)
  Day 14 DBP, 1 hour, n=23, 24 | 0.4 (4.18) | 0.0 (2.30)
  Day 14 DBP, 2 hours, n=23, 24 | 1.3 (3.75) | 0.4 (3.19)
  Day 14 DBP, 4 hours, n=23, 24 | 1.1 (4.17) | 1.1 (3.35)
  Day 14 DBP, 8 hours, n=23, 24 | 1.4 (3.27) | -0.2 (3.02)

14. Primary Outcome: Change From Baseline in Heart Rate at Day1 and Day 14 of the Respective Treatment Period
Description: Heart rate (HR) was measured at Day 1 and Day 14 of the respective treatment period. hr=hour. Baseline is defined as the pre-dose measurement at Day 1. Change from Baseline was calculated as the Day 14 value minus the Baseline value. Treatment, period, day (1 and 14), participant Baseline, period Baseline, and treatment*day interaction were fitted as fixed effects, and participant was fitted as a random effect.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Beats per minute
  Day 1, n=25, 25 | 84.4 (1.63) | 88.6 (1.63)
  Day 14, n=23, 24 | 89.4 (1.71) | 85.7 (1.67)
Statistical Analysis 1: Comparison: FF 100 µg/VI 25 µg vs FF 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-8.8 to 0.4] — Day 1 HR. The estimated value represents the treatment difference: FF/VI 100/25 µg minus FF 100 µg
Statistical Analysis 2: Comparison: FF 100 µg/VI 25 µg vs FF 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-1.1 to 8.5] — Day 14 HR. The estimated value represents the treatment difference: FF/VI 100/25 µg minus FF 100 µg

15. Primary Outcome: Maximum QTcF at Day 1 and Day 14 of the Respective Treatment Period
Description: QTcF is the QT domain corrected for heart rate by Fridericia's formula. Treatment, period, day (1 and 14), participant Baseline, period Baseline, and treatment*day interaction were fitted as fixed effects, and participant was fitted as a random effect.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
milliseconds
  Day 1 QTcF, n=25, 25 | 403.3 (1.98) | 402.2 (1.98)
  Day 14 QTcF, n=23, 24 | 404.0 (2.06) | 404.2 (2.02)
Statistical Analysis 1: Comparison: FF 100 µg/VI 25 µg vs FF 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-4.4 to 6.7] — Day 1 QTcF. The estimated value represents the treatment difference: FF/VI 100/25 µg minus FF 100 µg
Statistical Analysis 2: Comparison: FF 100 µg/VI 25 µg vs FF 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-6.0 to 5.5] — Day 14 QTcF. The estimated value represents the treatment difference: FF/VI 100/25 µg minus FF 100 µg

16. Secondary Outcome: AUC(0-t) and AUC(0-4) of FF on Day 14 of the Respective Treatment Period
Description: Area under the concentration-time (AUC) curve from time zero (pre-dose) to the last time AUC(0-t) and from time zero to 4 hours AUC(0-4) of quantifiable concentration of FF on Day 14 of the respective treatment period was measured. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PK Population.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: FF Pharmacokinetic (PK) Population: participants in the All Subjects Population for whom a PK sample was obtained and analyzed for FF.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms*hour per milliliter (pg*hr/mL)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 24 | 24
picograms*hour per milliliter (pg*hr/mL)
  AUC(0-t), n=23, 24 | 38.895 [21.630 to 69.941] | 32.880 [18.268 to 59.179]
  AUC(0-4), n=17, 15 | 86.14 [70.03 to 105.96] | 83.83 [71.49 to 98.30]

17. Secondary Outcome: Cmax of FF on Day 14 of the Respective Treatment Period
Description: Cmax is defined as the maximum observed concentration of FF on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: FF PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 23 | 24
picograms per milliliter (pg/mL) | 20.73 [15.16 to 28.36] | 21.16 [14.91 to 30.02]

18. Secondary Outcome: Tmax and Tlast of FF on Day 14 of the Respective Treatment Period
Description: tmax is defined as the time to reach the observed maximum concentration, and tlast is defined as the time of the last observed quantifiable concentration on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: FF PK Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Median (Full Range); unit: hours
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 24 | 24
hours
  tmax, n=20, 19 | 0.965 [0.00 to 2.07] | 0.500 [0.00 to 3.95]
  tlast, n=20, 19 | 4.030 [0.52 to 4.13] | 4.020 [1.03 to 4.05]

19. Secondary Outcome: AUC(0-t) and AUC(0-4) of VI on Day 14 of the Respective Treatment Period
Description: Area under the concentration-time (AUC) curve from time zero (pre-dose) to the last time AUC(0-t) and from time zero to 4 hours AUC(0-4) of quantifiable concentration of VI on Day 14 of the respective treatment period was measured. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the VI PK Population.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: VI PK Population: participants in the All Subjects Population for whom a PK sample was obtained and analyzed for VI.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms*hour per milliliter (pg*hr/mL)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 23 | 0
picograms*hour per milliliter (pg*hr/mL)
  AUC(0-t), n=23 | 44.297 [26.996 to 72.688] |
  AUC(0-4), n=11 | 119.19 [102.41 to 138.73] |

20. Secondary Outcome: Cmax of VI on Day 14 of the Respective Treatment Period
Description: Cmax is defined as the maximum observed concentration of VI on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: Participants received FF 100 µg in one of the two 14-day treatment periods. FF 100 µg was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 23 | 0
picograms per milliliter (pg/mL) | 44.21 [27.65 to 70.70] |

21. Secondary Outcome: Tmax and Tlast of VI on Day 1 of the Respective Treatment Period
Description: tmax is defined as the time to reach the observed maximum VI concentration, and tlast is defined as the time of the last observed quantifiable VI concentration on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: VI PK Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the VI PK Population.
Measure: Median (Full Range); unit: hours
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 23 | 0
hours
  tmax, n=21 | 0.170 [0.00 to 2.08] |
  tlast, n=21 | 3.870 [0.50 to 4.13] |

22. Secondary Outcome: Blood Glucose and Potassium Values on Day 14 of the Respective Treatment Period
Description: Blood glucose and potassium values were measured on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, and 4 hours post-dose. Weighted means were derived using the linear trapezoidal rule. Actual relative times were used for the calculation except where actual times were missing. If any actual times were missing, planned relative time were used for these observations. Treatment and period were fitted as fixed effects and participant was fitted as a random effect.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimoles per liter (mmol/L)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Millimoles per liter (mmol/L)
  Glucose, n=22, 24 | 5.578 (0.1495) [5.275 to 5.881] | 5.074 (0.1443) [4.781 to 5.367]
  Potassium, n=21, 23 | 4.059 (0.0448) [3.969 to 4.150] | 4.148 (0.0426) [4.062 to 4.234]

23. Secondary Outcome: Serum Cortisol (SC) Weighted Mean (0-12 Hours) on Day 14 of the Respective Treatment Period
Description: SC weighted mean was determined for each participant over the time period of 0-12 hours on Day 14 of the respective treatment period. SC weighted mean was derived by dividing the area under the concentration-time curve (AUC; defined as thearea under the concentration-time curve from time zero up to 24 hours) by the sample collection time interval. The sample collection time interval is defined as the difference between the time of the last cortisol sample and the time of the first cortisol sample. Samples were collected at the following time points: 0 (first blood draw/pre-dose); 2, 4, 8, and 12 hours (relative to the "0" time point). Weighted means were derived using the linear trapezoidal rule. Actual relative times were used for the calculation except where actual times were missing. If any actual times were missing, planned relative time were used for these observations. Treatment and period were fitted as fixed effects and participant was fitted as a random effect.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: nanomoles per Liter
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 23 | 23
nanomoles per Liter | 193.77 (0.069) [168.42 to 222.93] | 192.50 (0.069) [167.32 to 221.48]

24. Secondary Outcome: Average Oropharyngeal Cross-sectional Area on Day 1 and Day 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for the study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Pharyngometry data were recorded for each day (Day 1 and Day 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day X)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
centimeters squared (cm^2)
  Day 1, n=23, 23 | 4.13 (2.010) | 3.85 (2.043)
  Day 14, n=23, 23 | 3.76 (2.195) | 3.70 (2.279)

25. Secondary Outcome: Distance of Assessment on Day 1 and Day 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Distance of assessment is defined as the distance (length measured in centimeters [cm]) estimated to be from the lips to the larynx. Pharyngometry data were recorded for each day (Days 1 and 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
centimeters (cm)
  Day 1, n=23, 23 | 19.20 (1.097) | 19.24 (0.959)
  Day 14, n=23, 23 | 19.26 (0.717) | 19.10 (1.003)

26. Secondary Outcome: Oropharyngeal Volume on Day 1 and Day 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Oropharyngeal volume is defined as the volume (cm^3) of the mouth and throat estimated to be from the lips to the larynx. Pharyngometry data were recorded for each day (Days 1 and 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Liters per minute (L/min)
  Day 1, n=23, 23 | 79.49 (43.398) | 75.54 (44.195)
  Day 14, n=23, 23 | 72.35 (42.437) | 71.47 (45.841)

27. Secondary Outcome: Average Flow Rate and Peak Inspiratory Flow Rate (PIFR) on Day 1 and Day 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Average flow rate is defined as the average inspiratory flow rate (Liters [L]/min) across the inhalation profile when inhaling across the resistance of the inhaler. PIFR is defined as the Peak Inspiratory Flow Rate (L/min) of the inhalation profile when inhaling across the resistance of the inhaler.The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the average flow rate and PIFR were determined.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Liters per minute (L/min)
  Day 1, Average flow rate, n=23, 23 | 41.11 (11.294) | 42.72 (11.593)
  Day 14, Average flow rate, n=23, 23 | 42.29 (10.895) | 41.36 (10.354)
  Day 1, PIFR, n=23, 23 | 65.85 (16.649) | 67.60 (16.097)
  Day 14, PIFR, n=23, 23 | 67.36 (16.432) | 64.79 (15.886)

28. Secondary Outcome: Inhalation Time on Days 1 and 14 of of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Inhalation time is defined as the duration of the inhalation(s) when inhaling across the resistance of the inhaler. The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the inhalation time was determined.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Seconds (sec)
  Day 1, n=23, 23 | 0.97 (0.350) | 0.83 (0.385)
  Day 14, n=23, 23 | 0.96 (0.314) | 0.91 (0.347)

29. Secondary Outcome: Inhaled Volume on Days 1 and 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Inhaled volume is defined as the volume of air (Liters) inhaled during the inhalation across the resistance of the inhaler.
  The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the inhalaled volume was determined.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Liters
  Day 1, n=23, 23 | 0.69 (0.337) | 0.58 (0.285)
  Day 14, n=23, 23 | 0.68 (0.308) | 0.65 (0.352)

30. Secondary Outcome: Peak Pressure Drop on Days 1 and 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Peak pressure drop is defined as the maximum pressure drop (kilopascal [kPa]) achieved during inhalation across the resistance of the inhaler. The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was calculated for each day (Days 1 and 14 of the respective treatment period), and used for subsequent modeling and prediction of dose emission attributes.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Kilopascal (kpa)
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
Kilopascal (kpa)
  Day 1, n=23, 23 | 3.79 (1.706) | 3.97 (1.787)
  Day 14, n=23, 23 | 3.93 (1.877) | 3.67 (1.611)

31. Secondary Outcome: Total Emitted Dose (TED) on Day 14 of the Respective Treatment Period
Description: The total emitted dose (TED) is defined as the mass (micrograms) of the nominal dose that passes beyond the throat. The recorded inhalation profiles of the participants and the mouth-throat (oropharyngeal) models of the sizes that approximated to pharyngometry measurements of the participants were used in conjunction with the electronic Lung (eLung) for in vitro assessment. The eLung is a breathing simulator that replicates the selected inhalation profile with an active inhaler placed at the lips end of the selected ororpharyngeal model. After the dose is emitted from the inhaler, the analysis and assay of throat deposition and material passing beyond the throat was used to derive the nominal, minimum, and maximum predicted total emitted dose.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
micrograms
  Nominal TED FF, n=23, 23 | 87.58 (0.305) | 86.33 (1.505)
  Minimum TED FF, n=23, 23 | 87.64 (0.330) | 86.72 (1.589)
  Maximum TED FF, n=23, 23 | 87.51 (0.289) | 85.93 (1.534)
  Nominal TED VI, n=23, 0 | 20.26 (0.162) | NA (NA) — The TED of VI was not assessed in participants receiving only FF.
  Minimum TED VI, n=23, 0 | 20.22 (0.153) | NA (NA) — The TED of VI was not assessed in participants receiving only FF.
  Maximum TED VI, n=23, 0 | 20.29 (0.175) | NA (NA) — The TED of VI was not assessed in participants receiving only FF.

32. Secondary Outcome: Ex-throat Dose (ETD) and ETD <2 Microns on Day 14 of the Respective Treatment Period
Description: The ex-throat dose (ETD) and the "nominal ETD" is the mass (micrograms) of active investigational material that passes beyond the throat, nominal being the mean. The recorded inhalation profiles of the participants and the mouth-throat (oropharyngeal) models of the sizes that approximated to pharyngometry measurements of the participants were used in conjunction with the electronic Lung (eLung) for in vitro assessment. The eLung is a breathing simulator that replicates the selected inhalation profile with an active inhaler placed at the lips end of the selected ororpharyngeal model. After the dose is emitted from the inhaler, the analysis and assay of throat deposition and material passing beyond the throat was used to derive the nominal, minimum, and maximum predicted ETD and ETD <2 microns.
Time Frame: Day 14 of the respective treatment period (up to Study Day 63)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Number analyzed (Participants) | 25 | 25
micrograms
  Nominal ETD FF, n=23, 23 | 24.96 (5.801) | 24.34 (8.574)
  Minimum ETD FF, n=23, 23 | 23.38 (7.023) | 22.99 (9.120)
  Maximum ETD FF, n=23, 23 | 26.24 (4.825) | 25.48 (8.197)
  ETD <2 microns FF, n=23, 23 | 6.66 (0.948) | 5.97 (1.382)
  Minimum ETD <2 microns FF, n=23, 23 | 6.45 (0.788) | 5.77 (1.319)
  Maximum ETD <2 microns FF, n=23, 23 | 6.92 (1.147) | 6.21 (1.476)
  Nominal ETD VI, n=23, 0 | 8.54 (0.953) | NA (NA) — The ETD of VI was not assessed in participants receiving only FF.
  Minimum ETD VI, n=23, 0 | 8.33 (0.793) | NA (NA) — The ETD of VI was not assessed in participants receiving only FF.
  Maximum ETD VI, n=23, 0 | 8.80 (1.154) | NA (NA) — The ETD of VI was not assessed in participants receiving only FF.
  ETD <2 microns VI, n=23, 0 | 4.86 (1.162) | NA (NA) — The ETD of VI was not assessed in participants receiving only FF.
  Minimum ETD <2 microns VI, n=23, 0 | 4.60 (0.965) | NA (NA) — The ETD of VI was not assessed in participants receiving only FF.
  Maximum ETD <2 microns VI, n=23, 0 | 5.18 (1.409) | NA (NA) — The ETD of VI was not assessed in participants receiving only FF.

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the All Subjects Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | FF 100 µg/VI 25 µg | FF 100 µg
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg/VI 25 µg (N=25) | FF 100 µg (N=25)
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.